CLINICAL TRIAL: NCT00037544
Title: An Open-Label Study to Characterize the Safety and Efficacy of BDDrFVIII Manufactured by the Albumin Free Process (ReFacto AF) in the Treatment of Previously Treated Patients (PTP) With Severe Hemophilia A
Brief Title: Study Evaluating ReFacto AF in Severe Hemophilia A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Purpose: Treatment
Other Study IDs: 3082B1-306
Record Dates: First submitted 2002-05-17; First posted 2002-05-20 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Hemophilia A
Keywords: Severe; Hemophilia; A
MeSH Terms: conditions — Hemophilia A; Lymphoma, Follicular | interventions — Factor VIII

INTERVENTIONS:
Drug: ReFacto AF

SUMMARY:
To characterize the safety and efficacy of ReFacto AF in treating acute bleeding episodes during prophylaxis treatment, including neoantigenicity.

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia A (FVIII:C less than or equal to 2% at local laboratory)
* Previously treated patients with greater than or equal to 250 exposure days to any Factor VIII product
* Age greater than or equal to 12 years
* History of prophylaxis dosing at least twice per week on any Factor VIII product for at least 3 consecutive months within the 2 years prior to study enrollment unless the patient completed the previous pharmacokinetic study
* Adequate laboratory results

Exclusion Criteria:

* Presence of any bleeding disorder in addition to hemophilia A
* Concomitant therapy with immunosuppressive drugs
* Current or historical Factor VIII inhibitor
* Treatment with any investigational drug or device within the past 30 days

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer